CLINICAL TRIAL: NCT03279874
Title: Qualitative Interview Study Regarding Dentists' Repair Behaviour
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, PD Dr. med. dent., Dr. rer. medic., Senior Dental Practitioner, University Medical Center Goettingen
Other Study IDs: Interview-Repair; 22/9/17 (Other: Local Ethics Commission)
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Behavior
Keywords: decision-making; repair behavior; interviews
MeSH Terms: conditions — Behavior | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- German dentists: Dentists who are working in dental offices in Germany
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — Semi-structured one-on-one interviews

SUMMARY:
The aim of the present study is to determine dentists' barriers and facilitators for performing repairs on partially defective dental restorations.

DETAILED DESCRIPTION:
Potential barriers and facilitators for treating partially defective dental restorations by repair instead of complete replacement are going to be assessed by interviewing German dentists.

ELIGIBILITY:
Inclusion Criteria:

* Dentists who are working in dental offices in Germany and who are able to give written consent

Exclusion Criteria:

* Non-fulfillment of the inclusion criteria
* Lack of capacity to consent
* No German language skills in written and spoken language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dentists who are working in dental offices in Germany
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Completion of a questionnaire | 5 minutes
Interview | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kanzow, PD Dr. Dr. med. dent., M.Sc., Principal Investigator — Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany
Locations (1):
- University Medical Center Göttingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanzow P, Hoffmann R, Tschammler C, Kruppa J, Rodig T, Wiegand A. Attitudes, practice, and experience of German dentists regarding repair restorations. Clin Oral Investig. 2017 May;21(4):1087-1093. doi: 10.1007/s00784-016-1859-3. Epub 2016 Jun 2. PMID 27255959
- [Background] Kanzow P, Dieckmann P, Hausdorfer T, Attin T, Wiegand A, Wegehaupt FJ. Repair restorations: Questionnaire survey among dentists in the Canton of Zurich, Switzerland. Swiss Dent J. 2017 Apr 10;127(4):300-311. doi: 10.61872/sdj-2017-04-267. English, German. PMID 28480953
- [Background] Kanzow P, Wiegand A, Schwendicke F. Cost-effectiveness of repairing versus replacing composite or amalgam restorations. J Dent. 2016 Nov;54:41-47. doi: 10.1016/j.jdent.2016.08.008. Epub 2016 Aug 26. PMID 27575986
- [Result] Kanzow P, Kanzow AF, Wiegand A, Schwendicke F. Implementation of repairs in dental practice: Randomized behavior simulation trial. J Am Dent Assoc. 2023 Jul;154(7):610-619.e11. doi: 10.1016/j.adaj.2023.04.007. Epub 2023 May 22. PMID 37212760